CLINICAL TRIAL: NCT04253197
Title: Efficacy of Ultrasound Staging System in Prediction of Morbidly Adherent Placenta
Brief Title: Ultrasound Staging in the Placenta Accreta
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Nesreen Abdel Fattah Abdullah Shehata, Associate Professor in Obstetrics and Gynecology Department, Beni-Suef University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Beni-Suef 3-2017
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Obstetric Labor Complications; Staging of Placental Invasion
MeSH Terms: conditions — Obstetric Labor Complications | interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: Pregnant women in 3rd trimester
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Morbidly adherent placenta (Other): This arm was given stage according to ultrasound features.
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Pregnant women in 3rd trimester with anterior placenta previa and lower cesarean section scar. Ultrasound was done and according to parameters of the morbidly adherent placenta, a staging system was conducted.

SUMMARY:
The investigators evaluated the efficacy of a staging system introduced by the American Institute of ultrasound in medicine 2015 including sonographic parameters associated with morbidly adherent placenta for antenatal prediction of placental invasion.

DETAILED DESCRIPTION:
Morbidly adherent placenta (MAP) defines a spectrum of conditions, including placenta accreta, increta, and percreta, which are associated with significant maternal and fetal morbidity and mortality. Ultrasound evaluation, with grayscale, is the recommended first-line modality for diagnosing MAP. Grayscale ultrasound features suggestive of placenta accreta include the loss of myometrial interface or retroplacental clear space, reduced myometrial thickness and the presence of intraplacental lacunae. Using a staging system by antenatal ultrasound can predict placental invasion antenatally.

ELIGIBILITY:
Inclusion Criteria:

* Prior lower segment cesarean section
* Low lying anterior placenta
* Singleton pregnancy

Exclusion Criteria:

* Medical disorders
* vasa previa

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2019-12-25 (Actual)

PRIMARY OUTCOMES:
Confirmation of the stage of myometrial placental invasion | 1 hour
  By ultrasound, placental invasion in myometrium was given a stage

SECONDARY OUTCOMES:
Blood loss | 1 hour
  Documentation of complications intraoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-Suef University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albayrak M, Ozdemir I, Koc O, Demiraran Y. Post-partum haemorrhage from the lower uterine segment secondary to placenta praevia/accreta: successful conservative management with Foley balloon tamponade. Aust N Z J Obstet Gynaecol. 2011 Aug;51(4):377-80. doi: 10.1111/j.1479-828X.2011.01309.x. Epub 2011 Apr 18. PMID 21806571
- [Background] American institute of ultrasound in medicine 2015.